CLINICAL TRIAL: NCT05318404
Title: Comparison of Clinical Outcomes and Nutritional Status Between Conventional Oral Intake and Delayed Oral Intake With Jejunostomy Feeding After Esophagectomy: An Open Labeled Randomized Controlled Trial
Brief Title: Conventional Oral Intake vs Delayed Oral Intake With Jejunostomy Feeding After Esophagectomy (JNS Study)
Acronym: JNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1756
Record Dates: First submitted 2022-03-22; First posted 2022-04-08 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Esophageal Cancer; Surgery; Jejunostomy; Complications; Nutrition Related Cancer
Keywords: esophagectomy; esophageal cancer; nutritional support; jejunostomy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventinal feeding group (No Intervention): Start oral feeding 5-7 days after esophagectomy and discharge with soft blended diet as major energy source
- Delayed feeding group (Experimental): Start clear liquid fluid diet 5-7 days after esophagectomy and discharge with jejunostomy feeding as the major energy source. Start oral feeding at postoperative 1st visit
  Interventions: Dietary Supplement: Jejunostomy feeding

INTERVENTIONS:
Dietary Supplement: Jejunostomy feeding — Maintain jejunostomy feeding till postoperative 1st visit after esophagectomy in delayed feeding group
  Arms: Delayed feeding group

SUMMARY:
Comparison of nutritional and early surgical outcome between early and delayed oral feeding after esophagectomy for esophageal cancer

DETAILED DESCRIPTION:
Esophageal cancer is a highly aggressive malignancy that metastasizes to the lymph nodes and is associated with a poor prognosis. The 5-year overall survival rate is 40.0 % and the 30-day mortality rate is 1.7 %. Surgical resection is the most effective treatment for localized esophageal cancer; however, esophagectomy is extremely invasive and is associated with high morbidity and mortality rates.

Nutrition is one of the most important factors to consider after esophagectomy in order to reduce surgical mortality. The European Society for Parenteral and Enteral Nutrition guidelines recommend early tube feeding after major gastrointestinal surgery for cancer. Several studies have shown that enteral nutrition is more effective than parenteral nutrition in reducing postoperative complications in postesophagectomy patients. It has been reported that 5 to 7 days are required for anastomosis site healing. Therefore, many centers start oral feeding after esophagectomy on postoperative 7 days after anastomosis site evaluation, and enteral feeding via jejunostomy are maintained for nutritional support. However, the optimal timing for oral feeding after esophagectomy is still under debate.

In our center, the investigators routinely place jejunostomy tube for sufficient enteral feeding after esophagectomy. Before 2014, the investigators started oral feeding 5 to 7 days after esophagectomy and patients were discharged with soft blended diet. After 2014, the investigators changed our postoperative management protocols: 1) the investigators started only liquid diet 5 to 7 days after esophagectomy and maintained this feeding regimen until the first postoperative clinic visit with supplement of enteral feeding by jejunostomy tube. However, no studies have been conducted showing the optimal timing for oral feeding for esophagectomy patients for nutritional support and postoperative care.

The investigators hypothesized that delayed oral feeding after esophagectomy with jejunostomy feeding is superior to conventional oral feeding for nutritional support and early clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients who planned to undergo esophagectomy with esophageal reconstruction for esophageal cancer for curative purpose
* Patients who can understand the purpose and protocol of the clinical trial

Exclusion Criteria:

* BMI < 18kg/m2 or BMI > 25kg/m2
* Patients who needs colon of jejunum for esophageal reconstruction
* Patients who needed enteral feeding before esophagectomy
* Preoperative major organ failure (ex. renal failure requiring renal replacement, hepatic failure)
* Severe metabolic disorder (ex. uncontrolled diabetes mellitus, uncontrolled thyroid disease)
* Other patients who are not suitable for clinical trial

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Percentage of body weight loss | at postoperative 1st visit (postoperative 4-5 weeks)
  Percentage of body weight loss from preoperative body weight

SECONDARY OUTCOMES:
Postoperative complication rate | From date of randomization until the date of discharge after operation, assessed up to 2 months
  Postoperative complication rate
Complication related to jejunostomy feeding | From date of randomization until the date of discharge after operation, assessed up to 2 months
  Complication related to jejunostomy feeding
Postoperative Nutritional index | at postoperative 1st visit (postoperative 4-5 weeks), at postoperative 3-4 months
  GLIM criteria for malnutrition, handgrip strength, serum albumin, serum prealbumin
Postoperative daily total calorie intake | at postoperative 1st visit (postoperative 4-5 weeks), at postoperative 3-4 months
  Postoperative daily total calorie intake (kcal/day)
Postoperative daily protein intake | at postoperative 1st visit (postoperative 4-5 weeks), at postoperative 3-4 months
  Postoperative daily protein intake (g/day)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided